CLINICAL TRIAL: NCT01775670
Title: Off-the-Shelf Splints Versus Occupational Therapy Splints for Treatment of Trapeziometacarpal Arthrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the principal investigator leaving the institution and slow enrollment, we have decided to close the study prior to study completion
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2013-01-22; First posted 2013-01-25 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Trapeziometacarpal (TMC) Arthrosis
Keywords: Arthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Off-the-Shelf Splint (Experimental): Subjects in this arm will be managed with off-the-shelf splints for TMC arthrosis.
  Interventions: Device: Off-the-shelf splint
- OT Splint (Active Comparator): Subjects in this arm will be managed with a custom-made splint made by the Massachusetts General Hospital Occupational Therapists.
  Interventions: Device: OT Splint

INTERVENTIONS:
Device: Off-the-shelf splint — Subjects will use an off-the-shelf splint
  Arms: Off-the-Shelf Splint
Device: OT Splint — Subjects will use a splint custom-made by Massachusetts General Hospital Occupational Therapists.
  Arms: OT Splint

SUMMARY:
The specific aim is to compare the effectiveness of Off-the-Shelf splints and splints provided by Occupational Therapy for treatment of trapeziometacarpal (TMC) arthrosis.

DETAILED DESCRIPTION:
Trapeziometacarpal (TMC) arthrosis is so common, particularly in women, that it should be considered a normal part of the aging process. Overall radiographic prevalence of TMC arthrosis has been described to be as high as 91% in patients older than eighty years of age. It increases steadily from the age of 41 years, more rapidly in women than in men. Another study, conducted in the Netherlands, showed that in a population of 55 years and older, 67% of women and 55% of men had radiographic signs of arthrosis of the hand. It also found that the distal interphalangeal (DIP) joints are most commonly affected (47%), followed by the TMC joint (36%). However, it has been reported that in symptomatic arthrosis, TMC arthrosis contributes more to pain and disability than arthrosis of the interphalangeal joints. Psychosocial factors have been recognized as the strongest determinants of highly variable pain intensity and arm-specific disability. The pathophysiologic and psychosocial differences between patients who present to the doctor for treatment and those who do not are incompletely understood.

A hand-based thumb spica splint with the interphalangeal (IP) joint free is a specific nonoperative palliative treatment for TMC arthrosis. The goals of splint wear are improved comfort and function. The data regarding specific splint materials are limited, but suggest that shorter more flexible splints are preferred by patients and equally effective. Recently, the investigators looked into if there was a difference between thermoplast and neoprene hand-based thumb spica splints for treatment of TMC arthrosis. The neoprene splint was rated more comfortable than the thermoplast splint but otherwise there was no difference.

To the investigators' knowledge no studies have looked at the added value of occupational therapy in splint treatment for TMC arthrosis. The investigators believe that the time spent by occupational therapists (OTs) coaching patients on adaptive and palliative measures is valuable in addition to their technical skills but the investigators cannot draw any conclusions until the investigators research this in a prospective trial.

The investigators propose a two arm unblinded, randomized (1:1) controlled trial to evaluate if there is a difference between prefabricated off-the-shelf splints and splints provided by an OT with standard care coaching. The investigators want to determine if there is a difference in arm-specific disability, average pain, and satisfaction at an average of 2 months between splints provided by an OT and prefabricated off-the-shelf splints.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years of age and older
2. Clinical or radiological diagnosis of TMC arthrosis by MD
3. English fluency and literacy

Exclusion Criteria:

1. Prior surgical treatment of TMC arthrosis on same side
2. Prior treatment of TMC arthrosis on same side with a splint during the last two months
3. Prior injury of the trapeziometacarpal joint
4. Rheumatoid arthritis
5. Pregnant women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Off-the-Shelf Splint: Subjects in this arm will be managed with off-the-shelf splints for trapeziometacarpal (TMC) arthrosis.
  Off-the-shelf splint: Subjects will use an off-the-shelf splint
- OT Splint: Subjects in this arm will be managed with a custom-made splint made by the Massachusetts General Hospital (MGH) Occupational Therapists.
  Occupational Therapy (OT) Splint: Subjects will use a splint custom-made by MGH Occupational Therapists.
Period: Overall Study
Arm/Group | Off-the-Shelf Splint | OT Splint
Started | 1 | 3
Completed | 0 | 2
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- OT Splint: Subjects in this arm will be managed with a custom-made splint made by the MGH Occupational Therapists.
  OT Splint: Subjects will use a splint custom-made by MGH Occupational Therapists.
- Total: Total of all reporting groups
Arm/Group | Off-the-Shelf Splint | OT Splint | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (NA) — There is only one participant in this study arm. | 66.3 (4.2) | 64.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Disabilities of the Arm, Shoulder and Hand Quick Questionnaire (Quick-DASH)
Description: The short form of the Disabilities of Arm Shoulder and Hand to assess upper extremity disability. The scale range is from 0-100, where 0 is no difficulty performing tasks and 100 is the most difficulty or unable to complete any tasks.
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 1 | 2
units on a scale | 4.5 (NA) — There was only one participant's data available therefore no standard deviation calculated. | 29.5 (6.43)

2. Primary Outcome: Change From the Baseline in the Disabilities of the Arm, Shoulder and Hand Quick Questionnaire (Quick-DASH) at 2 Months After Enrollment
Description: The short form of the Disabilities of Arm Shoulder and Hand to assess upper extremity disability. The scale range is from 0-100, where 0 is no difficulty performing tasks and 100 is the most difficulty or unable to complete any tasks. This was measured 2-month after treatment.
Time Frame: 2 months after enrollment
Population: The one subject in the off-the-shelf group was lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
units on a scale |  | 20.5 (6.85)

3. Primary Outcome: Thumb Pain at Enrollment
Description: 11-point ordinal pain scale to assess the amount of pain. The scale range is from 0-10, where 0 is no pain at all and 10 is the worst pain ever had.
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 1 | 2
units on a scale | 3 (NA) — There was only one subject with data to analyze, therefore no standard deviation possible. | 5.5 (3.5)

4. Primary Outcome: Average Satisfaction With the Splint 2 Months After Enrollment
Description: Average satisfaction with splint treatment will be assessed 2 months after enrollment. 11-point ordinal pain scale to assess the amount of satisfaction. The scale range for satisfaction is from 0-10, where 0 is dissatisfaction and 10 is complete satisfaction with the splint.
Time Frame: At 2 months after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
units on a scale |  | 4 (1.4)

5. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) - Depression
Description: A computerized assessment of depression measured at enrollment. The average T score of the U.S. population is 50, so the T score reported compares the study population to the U.S. population, where a T score greater than 50 is worse than the average and a T score less than 50 is better than the average.
Time Frame: At Enrollment
Population: The data was not recorded for the 1 patient randomized to the off-the-shelf group.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
T score |  | 38.9 (6.6)

6. Secondary Outcome: PROMIS Pain - Interference
Description: A computerized assessment of pain interference measured at enrollment. The average T score of the U.S. population is 50, so the T score reported compares the study population to the U.S. population, where a T score greater than 50 is worse than the average and a T score less than 50 is better than the average.
Time Frame: At Enrollment
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
T score |  | 54.5 (2.33)

7. Secondary Outcome: Thumb Metacarpophalangeal (MCP) Joint in Resting Position (Degrees)
Description: Measurements of thumb metacarpophalangeal (MCP) joint in resting position.
Time Frame: At Enrollment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
degrees |  | 7.5 (3.5)

8. Secondary Outcome: Thumb MCP in Pinch Position (Degrees)
Description: Measurements of thumb MCP in pinch position.
Time Frame: At Enrollment
Population: The measurement of the thumb MCP joint in a pinch position was the same, 10 degrees, for the 2 subjects in the OT splint group, therefore the standard deviation is 0.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 2
degrees |  | 10 (0)

9. Secondary Outcome: Thumb Pinch Strength
Description: Measurement of thumb pinch strength using a pinch meter. Subjects place the pinch meter between their thumb and index finger and pinch down to record the pinch strength.
Time Frame: At Enrollment
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 1 | 2
pounds | 7.67 (NA) — There was only one subject's data available to analyze, therefore there is no standard deviation. | 10.67 (0.94)

10. Secondary Outcome: Thumb Grip Strength
Description: Grip strength of the affected hand was measured at enrollment using a dynamometer. The subject squeezes the handle of the dynamometer to maximum capability to measure grip strength. Each subject completed the grip strength measurement 3 times on the affected hand to get an average grip strength of the affected hand.
Time Frame: At Enrollment
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 1 | 2
pounds | 24.67 (NA) — There was only one subject's data available to analyze, therefore there is no standard deviation available to report. | 39.67 (14.61)

11. Primary Outcome: Average Pain 2 Months After Enrollment
Description: Average pain will be assessed 2 months after enrollment. 11-point ordinal pain scale to assess the amount of pain. The scale range for pain is from 0-10, where 0 is no pain and 10 is the worst pain.
Time Frame: At 2 months after enrollment
Population: Subjects did not complete the pain scale questionnaire at the follow up visit.
Arm/Group | Off-the-Shelf Splint | OT Splint
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Off-the-Shelf Splint | OT Splint
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes